CLINICAL TRIAL: NCT00003977
Title: A Phase I Study of Immunization With Alternating Human Papillomavirus E7 Lipopeptide Epitope Vaccine and Dendritic Cells Presenting the E7 Epitope for the Treatment of Recurrent or Persistent Cervical Cancer
Brief Title: Vaccine Therapy in Treating Patients With Recurrent or Persistent Cervical Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Steward St. Elizabeth's Medical Center of Boston, Inc. (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067180; SEMC-980016; NCI-T98-0072
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2009-02-09 (Estimated); Status verified 2003-12

CONDITIONS: Cervical Cancer
Keywords: stage III cervical cancer; recurrent cervical cancer; stage IB cervical cancer; stage IIB cervical cancer; stage IVB cervical cancer; stage IA cervical cancer; stage IIA cervical cancer; stage IVA cervical cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — oncogene protein E7, Human papillomavirus type 16

INTERVENTIONS:
Biological: human papillomavirus 16 E7 peptide
Procedure: in vitro-treated peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Vaccines may make the body build an immune response to kill tumor cells.

PURPOSE: Phase I trial to study the effectiveness of vaccine therapy in treating patients with recurrent or persistent cervical cancer that cannot be treated with surgery or radiation therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate alternating vaccination with lipidated human papillomavirus 16 E7 peptide (HPV-16 E7) and autologous dendritic cells pulsed with immunogenic HPV-16 E7 in terms of toxicity, immunologic reactivity, and therapeutic efficacy in patients with recurrent or persistent cervical cancer.

OUTLINE: This is a dose-escalation study of dendritic cell-human papillomavirus 16 E7 (HPV-16 E7) peptide vaccine.

Patients undergo leukapheresis to obtain peripheral blood mononuclear cells for activation to dendritic cells on days 0 and 28. Patients receive lipidated HPV-16 E7 peptide vaccine subcutaneously on days 1 and 14 and dendritic cell-HPV-16 E7 peptide vaccine IV over 15-30 minutes on days 7 and 21. Treatment continues in the absence of disease progression or unacceptable toxicity. Patients with stable disease or complete or partial response may receive one additional treatment course, beginning 6 weeks after the end of the first course.

Cohorts of 3-9 patients receive escalating doses of dendritic cell-HPV-16 E7 peptide vaccine. The maximum tolerated dose is defined as the dose preceding that at which 2 of 6 patients experience dose limiting toxicity.

A parallel cohort of patients receives dendritic cell-HPV-16 E7 peptide vaccine IV over 15-30 minutes on days 7 and 14, but does not receive lipidated HPV-16 E7 peptide.

Patients are followed at one week.

PROJECTED ACCRUAL: Approximately 27 patients will be accrued for this study at a rate of 15 patients per year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven recurrent or persistent cervical cancer not amenable to surgery or radiotherapy
* Measurable and evaluable disease
* HLA-A2 positive

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* More than 3 months

Hematopoietic:

* WBC greater than 3,000/mm^3
* Platelet count greater than 100,000/mm^3
* Hemoglobin greater than 8.0 g/dL
* No coagulation disorders

Hepatic:

* Bilirubin less than 2.0 mg/dL
* SGOT less than 4 times upper limit of normal

Renal:

* Creatinine less than 1.5 mg/dL OR
* Creatinine clearance greater than 75 mL/min

Cardiovascular:

* No major cardiovascular illness

Pulmonary:

* No major pulmonary illness

Other:

* HIV negative
* Hepatitis B surface antigen negative
* No active systemic infection
* Not pregnant
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least one month since prior biologic therapy

Chemotherapy:

* At least one month since prior chemotherapy

Endocrine therapy:

* At least one month since prior endocrine therapy
* No concurrent steroid therapy

Radiotherapy:

* See Disease Characteristics
* At least one month since prior radiotherapy

Surgery:

* See Disease Characteristics
* At least one month since prior surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-11

CONTACTS AND LOCATIONS:
Overall Officials: Michael A. Steller, MD, Study Chair — Steward St. Elizabeth's Medical Center of Boston, Inc.
Locations (1):
- St. Elizabeth's Medical Center, Boston, Massachusetts, United States